CLINICAL TRIAL: NCT01320566
Title: A Continuation Study of the AeriSeal® System Administered at 3 to 4 Sites During a Single Treatment Session for Lung Volume Reduction in Patients With Advanced Emphysema
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aeris Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-C10-003PLV
Record Dates: First submitted 2011-03-15; First posted 2011-03-22 (Estimated); Last update posted 2013-11-14 (Estimated); Status verified 2013-11

CONDITIONS: Pulmonary Emphysema; Chronic Obstructive Pulmonary Disease(COPD); Lung Diseases
Keywords: Polymeric Lung Volume Reduction (PLVR); Bolilogic Lung Volume Reduction (BLVR); AeriSeal; treatment; device; breathing; COPD; emphysema; heterogeneous; homogeneous; Pathologic Processes; Respiratory Tract Diseases; Lung Diseases; Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Emphysema; Pulmonary Disease, Chronic Obstructive; Lung Diseases; Respiratory Aspiration; Emphysema; Pathologic Processes; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AeriSeal System — Not applicable. Follow-Up study only.

SUMMARY:
The purpose of this study is to assess the long term safety and efficacy of AeriSeal System treatment administered at up to 4 subsegments during a single treatment session for lung volume reduction in patients with advanced emphysema through 48 weeks after treatment.

DETAILED DESCRIPTION:
Emphysema is a progressive, debilitating disease characterized by destruction of lung tissue as a result of inflammation caused by exposure to noxious inhaled agents for extended periods. The most common cause of this condition is cigarette smoking, although genetic, occupational, and environmental causes account for up to 10% of cases. Despite aggressive public health initiatives aimed at discouraging the use of cigarettes, smoking-related lung diseases remain a significant cause of disability and death worldwide. Due to the number of current and new smokers, emphysema is expected to remain a leading cause of morbidity and mortality for years to come.

The AeriSeal System is a novel device system being developed for the treatment of advanced emphysema. The AeriSeal System is administered bronchoscopically, and designed to provide the physiological benefits of lung volume reduction without the risks and cost of major surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been enrolled in the 03-C10-002PLV Aeris' Investigational Study and completed a minimum of 12 weeks of follow-up following AeriSeal System treatment.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Percent Volume of Lung | 48 Weeks following treatment
  Computed Tomography (CT) evidence of lobar volume reduction at site(s) of AeriSeal Foam Sealant administration at 48 weeks post treatment, assessed quantitatively by digital integration of CT dicom images collected using a standardized image acquisition and reconstruction algorithm.

SECONDARY OUTCOMES:
Change in the ratio of Residual Volume (RV) to Total Lung Capacity (TLC) | 24 and 48 weeks following treatment
  Change from baseline at 24 and 48 weeks in RV/TLC
Change in Forced Expiratory Volume in 1 Second (FEV1) | 24 and 48 weeks following treatment
  Change from baseline at 24 and 48 weeks in FEV1
Change in Forced Vital Capacity (FVC) | 24 and 48 weeks following treatment
  Change from baseline at 24 and 48 weeks in FVC
Change in distance walked in six minutes | 24 and 48 weeks following treatment
  Change from baseline at 24 and 48 weeks in 6 Minutes Walk Test (6MWT)
Change in Medical Research Council Dyspnea (MRCD) score | 24 and 48 weeks following treatment
  Change from baseline at 24 and 48 weeks in MRCD score
Change in St. George's Respiratory Questionnaire (SGRQ)domain score | 24 and 48 weeks following treatment
  Change from baseline at 24 and 48 weeks in SGRQ total domain score

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - The Soroka Medical Center, Beersheba
  - The Rabin Medical Center, Petah Tikva

REFERENCES:
- See also: Aeris Therapeutics — http://www.aerist.com/